CLINICAL TRIAL: NCT07353476
Title: Postoperative Involved-field Nodal Radiotherapy Plus Anti-PD-1 Maintenance Versus Anti-PD-1 Maintenance Alone in Patients With ypTanyN⁺M0 NSCLC After Neoadjuvant Chemoimmunotherapy and R0 Resection: A Single-center Randomized Phase II Study
Brief Title: Radiotherapy Plus Anti-PD-1 Versus Anti-PD-1 Alone in ypTanyN⁺M0 NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2026GRI
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); Post Surgical
Keywords: Radiotherapy; Adjuvant therapy; Lymph node
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Involved-field radiotherapy to regional draining lymph nodes + PD-1 maintenance (Active Comparator)
  Interventions: Radiation: radiotherapy; Drug: PD -1/PD-L1 monoclonal antibody
- No radiotherapy (standard of care) + PD-1 maintenance (Active Comparator)
  Interventions: Drug: PD -1/PD-L1 monoclonal antibody

INTERVENTIONS:
Radiation: radiotherapy — Postoperative external beam radiotherapy to regional draining lymph nodes (e.g., ipsilateral mediastinal and hilar nodal stations involved or at high risk), based on pre-treatment imaging and surgical/pathologic findings.
  Suggested dose: 50-54 Gy in 25-27 fractions (2.0-2.16 Gy per fraction, once daily, 5 days per week), delivered with 3D-CRT or IMRT per institutional standards.
  Arms: Involved-field radiotherapy to regional draining lymph nodes + PD-1 maintenance
Drug: PD -1/PD-L1 monoclonal antibody — Anti-PD-1 monoclonal antibody administered intravenously every 3 weeks for up to 1 year (or until disease recurrence, unacceptable toxicity, or withdrawal). The specific agent and dose will follow the neoadjuvant regimen and local regulatory approval.

SUMMARY:
Patients with stage III non-small-cell lung cancer (NSCLC) who receive neoadjuvant chemoimmunotherapy may achieve good response in the primary tumor but still have residual nodal disease after surgery (ypTanyN⁺M0), which is associated with poor prognosis in retrospective analyses from our center. In prior trials such as LungART and PORT-C, postoperative radiotherapy (PORT) did not improve disease-free survival in completely resected stage IIIA-N2 NSCLC after adjuvant chemotherapy, suggesting that PORT should not be used indiscriminately. However, recent preclinical and translational data indicate that radiotherapy can enhance antitumor immunity, remodel the tumor microenvironment, and synergize with immune checkpoint inhibitors via immunogenic cell death, improved T-cell trafficking, and tertiary lymphoid structure formation.

This single-center randomized phase II study will evaluate whether adding postoperative involved-field nodal radiotherapy to standard PD-1 maintenance therapy can improve disease-free survival compared with PD-1 maintenance alone in patients with ypTanyN⁺M0 NSCLC after neoadjuvant chemoimmunotherapy and R0 resection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, male or female.
* Histologically confirmed NSCLC (adenocarcinoma, squamous cell carcinoma, or other NSCLC subtypes).
* Clinical stage IIIA/IIIB at initial diagnosis, deemed suitable for neoadjuvant chemoimmunotherapy followed by surgery according to MDT.
* Completed 2-4 cycles of platinum-based doublet chemotherapy plus PD-1 inhibitor as neoadjuvant therapy.
* Underwent R0 resection (anatomical lobectomy or pneumonectomy with mediastinal lymph node dissection).
* Postoperative pathological stage ypT_anyN⁺M0 (residual nodal metastasis in mediastinal or hilar lymph nodes).
* ECOG performance status 0-1.
* Adequate hematologic, hepatic, and renal function per protocol-defined lab thresholds.
* Able to start postoperative radiotherapy and/or PD-1 maintenance within 4-10 weeks after surgery (or after recovery from postoperative complications, as clinically appropriate).
* Signed written informed consent.

Exclusion Criteria:

* Positive surgical margins (R1 or R2) or incomplete resection.
* Prior thoracic radiotherapy that would overlap with planned treatment fields.
* Active, uncontrolled infection or unresolved ≥ Grade 2 immune-related adverse events.
* History of severe autoimmune disease requiring systemic immunosuppression.
* Uncontrolled interstitial lung disease or significant pulmonary fibrosis.
* Symptomatic or untreated central nervous system metastases at enrollment.
* Any condition that, in the investigator's judgment, would compromise patient safety or protocol compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | 3 years
  Time from date of surgery to first documented recurrence (locoregional or distant) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Time from surgery to death from any cause (up to 5 years).
Incidence of Treatment-Emergent Adverse Events | Through treatment completion, an average of 1 year
  Incidence, type, and severity of adverse events graded by CTCAE v5.0, including radiation pneumonitis and immune-related toxicities.

IPD SHARING:
Plan to Share IPD: No